CLINICAL TRIAL: NCT07105332
Title: Investigation of a Sub-Conjunctival Insert
Brief Title: Feasibility Trial of a Sub-conjunctival Insert
Acronym: OMI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: terminated after the concept feasibility was succesfully proved, no safety issues
Sponsor: EyeSense GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: P-1.1-C-01
Record Dates: First submitted 2022-09-05; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-03

CONDITIONS: Diabetes (DM)
Keywords: sub-conjunctival implant; flash glucose monitoring; EyeSense, eye implant, glucose measurement in the eye
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort - Healthy subjects (Experimental): 2 healthy subjects will test OMI and Photometer for a period of up to 5 months: with sub-conjunctivaly implanted OMI participating on in-clinic sessions to optimize and adjust the measurement system (photometer).
  Interventions: Device: OMI and Photometer
- Cohort - Diabetic patients (Experimental): 8 diabetic patients will test OMI and Photometer: wearing sub-conjunctivaly implanted OMI for a period of up to 10 months and participating on up to 20 in-clinic sessions with blood glucose challenge to measure the performance of the system.
  Interventions: Device: OMI and Photometer

INTERVENTIONS:
Device: OMI and Photometer — A glucose sensitive ocular mini insert (OMI) is placed sub-conjunctivaly. When exited by photometer the glucose concentration is measured.

SUMMARY:
The purpose of this single-centre, open label prospective study is to investigate a novel ocular mini insert (OMI) for detection of blood glucose levels in human subjects. First, the optimal technical parameters for measurement are determined on healthy subjects. Secondly, performance measurements follow investigating relationship between OMI signal and blood glucose in diabetes patients during short sessions with oral glucose tolerace test.

ELIGIBILITY:
Inclusion Criteria:

1. Be of legal age or alternatively above 16 with written persmission of legal guardian.
2. Signed written Informed Consent.

Exclusion Criteria:

1. Pregnant or lactating females.
2. Poorly controlled diabetes mellitus with prior hemoglobin A1C greater than 10% or fasting glucose over 150 mg/dl.
3. Any known allergies, especially iodine.
4. Glaucoma patient.
5. Any acute disease.
6. Any present condition that would prevent from fasting or glucose challenge.
7. Any present condition that would prevent from insertion.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2006-12 (Actual); Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Correlation between OMI signal and blood glucose | 1-2 times weekly for 10 weeks after insertion
  Correlation between OMI fluorescence readings of subconjunctival interstitial fluid glucose concentration and capillary blood glucose level
Adverse Events Reporting | at each visit, up to 10 months
  wound healing and conjunctival hyperaemia

SECONDARY OUTCOMES:
Sensitivity and signal to noise ratio of the photometer | 1-2 times weekly for 10 weeks after insertion
Long term stability of insert | 1-2 times weekly for 10 weeks after insertion
  signal drift and stability of measurement
Targeting of measurement beam | 1-2 times weekly for 10 weeks after insertion
Subjective impressions | 10 months
  subjecs has to answer a questionnaire
Lag time | 1-2 times weekly for 10 weeks after insertion
  evaluation between device readings and blood glucose concentration

CONTACTS AND LOCATIONS:
Overall Officials: Holger Mietz, Prof. Dr., Principal Investigator — 63739 Aschaffenburg, Germany

IPD SHARING:
Plan to Share IPD: No